CLINICAL TRIAL: NCT03032328
Title: Comprehensive Assessment of Vascular and Autonomic Function in Children With Low Vitamin D
Brief Title: Vitamin D Deficiency and Dysautonomia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00036629
Record Dates: First submitted 2016-11-22; First posted 2017-01-26 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2022-04

CONDITIONS: Vitamin D Deficiency; Orthostatic Intolerance; Nausea
MeSH Terms: conditions — Vitamin D Deficiency; Orthostatic Intolerance; Nausea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vitamin D supplement (Experimental): patient's will be given a vitamin D
  Interventions: Dietary Supplement: vitamin D supplement

INTERVENTIONS:
Dietary Supplement: vitamin D supplement — Patients will be given a dose of vitamin D for at least 2 months

SUMMARY:
In previous work the investigator identified a group of children between the ages of 10-18 years whose diagnostic workup for chronic nausea unexplained by conventional diagnostic tests has unexpectedly revealed underlying cardiovascular instability manifesting as orthostatic intolerance, primary defined as postural orthostatic tachycardia syndrome (POTS) (88%). While this is an atypical initial presentation for orthostatic intolerance in general, the investigator believes that the cardiovascular problem is serious and represents a cause of the nausea in a majority of these individuals, as treatment of the POTS with fludrocortisone reduced the symptoms of nausea. While fludrocortisone treatment abrogates the fall in baroreflex sensitivity (BRS) during tilt in part, it did not completely correct the tachycardia symptoms or the BRS suppression during HUT. Furthermore it caused an elevation in MAP in supine position, which may lead to future cardiovascular problems such as early onset hypertension and cardiac hypertrophy. This argues for a different treatment approach. The investigator presents preliminary data in this application revealing that OI subjects tend to have lower 25-hydroxy vitamin D (25(OH)D) compared to non OI subjects.

DETAILED DESCRIPTION:
The investigators approach will combine HUT testing coupled with autonomic testing that includes continuous blood pressure and HR measurements, Baroreflex Sensitivity and Hear Rate Variability, to establish objective autonomic profiles, along with vascular testing including Pulse Wave Velocity, Ankle Brachial Index at rest and measures of blood volume of different compartments, Systemic Vascular Resistance and cardiac output at rest and in response to hand-grip stress. This will allow the treating physician to provide patients with a specific diagnosis, and ultimately develop data for more focused, rational treatments than currently achieved. The full vascular profile is also novel and has the potential to improve therapeutic management of the participants independent of the outcomes with the vitamin D supplementation. This study is designed to recruit 80 participants into 4 groups of 20 each. The 4 groups represent non OI (those recruited from the clinics for nausea but without a positive tilt test) or those showing orthostatic intolerance (POTS alone, OH, and syncope). The general objective of this proposal is to address this gap in knowledge by determining vascular function, the neurohumoral profile and autonomic status supine and in response to HUT in OI subjects with low vitamin D levels in comparison with subjects who test negative for OI on the HUT.

The investigators aim to examine the effect of vitamin D replacement on these measures, providing the possibility of therapeutic use of vitamin D to treat or ameliorate the symptoms associated with OI.

ELIGIBILITY:
Inclusion Criteria:

* The age range of 10-18 years was chosen as we anticipate these patients will be capable of adequately answering nausea symptom questionnaires and cooperating during autonomic and tilt table testing
* Patients will be recruited from the pediatric GI clinic if they meet Rome III criteria for childhood functional dyspepsia with nausea as the predominant symptom which includes: persistent or recurrent pain or discomfort (including nausea) in the upper abdomen not relieved with defecation and not associated an inflammatory, anatomic, metabolic, or neoplastic process
* Patients will be recruited from the pediatric cardiology clinic for presenting symptoms of unexplained syncope not associated with cardiac anatomic anomalies or other identified cardiac pathology

Exclusion Criteria:

* Patients will be excluded if a metabolic, mechanical, or mucosal inflammatory cause has been defined to explain their gastrointestinal symptoms. This would include, for example, a diagnosis of inflammatory bowel disease, celiac disease, liver or pancreatic disease, hiatal hernia, or bowel obstruction
* Patients with significant cardiac or cardiovascular disease, malignancy, or other comorbid conditions precluding successful completion of a 45 minute tilt test will be excluded.
* Subjects who are incapable or unwilling to discontinue medications affecting autonomic function will be excluded.
* Patients with diabetes will be excluded due to the possibility that the autonomic dysfunction results from a peripheral neuropathy. (We have successfully recruited these numbers of subjects in less than 2 years in a previous study of similar design
* Patients who are pregnant

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Improvement of orthostatic intolerance symptoms usint tilt table test | 2 months
  assessment of orthostatic intolerance will be done using tilt table test

SECONDARY OUTCOMES:
improvement of nausea symptoms | 2 months
  assessment of nausea symptoms will be done using nausea questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Shaltout, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT03032328/ICF_000.pdf